CLINICAL TRIAL: NCT02359786
Title: Retrospective Registry To Enhance the Understanding of the Variability, Progression and Treatment of Various Disorders
Brief Title: RAHM Foundation Retrospective Study of Various Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rahm Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RAHM 1002 v.6
Record Dates: First submitted 2015-01-29; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Pain, Spinal Surgeries, Hip and Knee Joint Replacement, Adverse Events
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Genetic Testing Subjects undergoing genetic testing
- Topicals Subjects using topical compounds
- Patients undergoing Spinal Surgery using IOM
- Spine Patients undergoing cervical or lumbar surgery
- Total Joint Patients undergoing knee and hip replacement
- UDT (unrinary drug test) Patients who are given a UDT

SUMMARY:
This is a retrospective data collection on treatment of various disorders. This registry will include a variety of different products, implants, technologies and procedures. The registry will also collect any adverse events/complications that occur during or following treatment of these conditions. The data may be utilized to develop strategic treatment pathways and/or benchmarking that will improve patient care. Ultimately, the goal of the registry is to enhance the understanding of healthcare and the treatment in these disease states.

DETAILED DESCRIPTION:
The purpose is to collect data on patients with a variety of disorders. This includes point of care (primary care, internal medicine, pain management providers, etc.) as well as a variety of specialty providers including neurosurgeons, orthopedic surgeons, oncologists, and dermatologists. The retrospective data collection will consist of a core set of data if available. The registry will attempt to collect data prior to surgery/treatment/procedures, during surgery, and various time points following surgery/treatment/procedures. The data will include, but is not limited to demographic data, past medical history, previous treatments, time off of work, type of surgery performed, products/implants/procedures/technology used during surgery, treatments/procedures/technology used for non-surgical conditions, anesthesia used during surgery, complications/adverse events following surgery and or treatment, outcome tools, imaging results, pain assessment, pain medication utilization, length of hospital stay, unplanned hospital admissions, revision surgery, adjacent level disease, genetic testing, urinary drug testing, other diagnostic or assessment testing, patient return to work and patient return to normal activity. The data collected will vary depending on disease state and treatment. This registry will also allow for comparisons on different treatments, procedures, etc. with a goal of developing the best pathways for a variety of different disease states.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet eligibility criteria across 1 of the 6 therapeutic areas

Exclusion Criteria:

* Subjects who do not meet eligibility criteria for any of the 6 therapeutic areas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with various disorders
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
sensory and motor deficits analysis, adverse events, changes in pain, changes in disability, return to work/usual activities, lenttgh of stays, hospital readmission rates, medication compliance rates | 60 months